CLINICAL TRIAL: NCT04617054
Title: A Phase II, Multicenter, Open, Basket Study of AB-106 to Treat the Subjects With Local Progression or Systemic Metastasis Solid Tumors With NTRK Gene Fusion
Brief Title: Phase II Study of AB-106 to Treat Patients With Solid Tumors With NTRK Gene Fusion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued early by the Sponsor for business reasons on 06 Dec 2024
Sponsor: Nuvation Bio Inc. (Industry)
Collaborators: AnHeart Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-106-C205
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm trial whereby all consented, enrolled, eligible patients receive AB-106 (Experimental)
  Interventions: Drug: AB-106

INTERVENTIONS:
Drug: AB-106 — 600mg QD for each subjects.

SUMMARY:
AB-106 will be administered once a day. Each treatment cycle is defined as 21 days of continuous medication. Dosing will continue until any of the following conditions are met: disease progression, intolerable drug-related adverse events, researchers recommend discontinuation of treatment, withdrawal of informed consent, pregnancy during the study, use of other anti-tumor therapy, loss of follow-up, death and other causes, whichever occurs first.

The study includes a screening period, treatment period, safety follow-up and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with locally advanced or metastatic solid tumors harboring NTRK1, NTRK2, or NTRK3 fusion genes (anticipated to translate into fusion proteins with a functional TrkA/B/C kinase domain);
2. Participants who had failed standard of care or refused standard of care;
3. Participants must have had at least 1 measurable lesion as defined by RECIST 1.1;
4. For participants diagnosed with a primary CNS tumor, the following criteria should have been met:

   * Must have received previous treatment, including radiotherapy (with clear progression before C1D1), chemotherapy, and targeted therapy (completed at least 4 weeks before C1D1).
   * At least 1 lesion must be measurable in two dimensions (confirmed by MRI and assessable as per RANO criteria), and each dimension of at least 1 measurable lesion must be ≥1 cm, and can be observed on more than 1 imaging slice.
5. Male or female participants ≥18 years old;
6. ECOG PS score of ≤1;
7. The Investigator judged that the participant's life expectancy was more than 3 months;
8. Within 7 days prior to enrollment, laboratory tests had to meet the following criteria (requiring no blood or blood product transfusion, no use of hematopoietic stimulants, or other medications to correct blood cells within 14 days prior to enrollment):

   * Absolute neutrophil count ≥1.5×109/L, platelets ≥80×109/L, and hemoglobin ≥90 g/L.
   * Serum AST and serum ALT ≤2.5×the upper limit of normal (ULN); AST and ALT ≤5×ULN for participants with liver tumors.
   * Total bilirubin ≤1.5×ULN. Participants with a known history of Gilbert's syndrome and an abnormal increase in indirect bilirubin are eligible.
   * Serum creatinine ≤2.0×ULN; urine dipstick for urine protein <2+; if ≥2+, a 24-hour urine protein should be quantified and total urine protein <1 g.
9. Coagulation: International normalized ratio (INR) ≤1.5, and partial prothrombin time or activated partial thromboplastin time (APTT) ≤1.5×ULN;
10. Participants must have been able to provide archived or newly obtained tumor tissue specimens (including consent for the collection of new biopsy specimens);
11. During the treatment period and for at least 90 days after completing study drug, participants agreed to use effective contraceptive measures (excluding males post-vasectomy, or females who were post-sterilization and postmenopausal). Women of childbearing potential were required to have a negative blood human chorionic gonadotropin (HCG) test within 7 days prior to the first dose;
12. Prior to enrollment, participants (or their legal representatives) had been fully informed and had signed and dated the informed consent form (ICF).

Exclusion Criteria:

1. Underwent treatment in another therapeutic clinical study within 4 weeks prior to the first dose of taletrectinib;
2. Participants who had suffered a cerebrovascular accident (excluding transient ischemic attacks) within 3 months before enrollment;
3. Participants with Grade ≥2 toxicity reactions from previous treatments which did not resolve, except for AEs deemed as not posing a safety risk (such as alopecia, neuropathy, and specific laboratory test abnormalities);
4. Participants with symptomatic or unstable brain metastases (participants with asymptomatic brain metastases may be eligible), and those with primary CNS tumors may be included if their condition was stable for at least 7 days;
5. Participants who underwent major surgery or radiotherapy within 28 days prior to enrollment (participants who received palliative radiotherapy for bone metastasis pain and brain metastasis radiotherapy within 2 weeks before enrollment were allowed to participate), or participants who were expected to require major surgery during the study;
6. Known interstitial lung disease, interstitial fibrosis, or pneumonitis induced by tyrosine kinase inhibitors;
7. Participants with active, uncontrollable systemic bacterial, viral, or fungal infections, or diseases such as diabetes or hypertension unmanageable with medication, or other systemic diseases that would hinder compliance with the study procedures;
8. Active hepatitis B or C infection (HBsAg positive and/or HBcAb positive with HBV DNA ≥104 copies or ≥2000 IU/mL; HCV antibody positive and HCV-RNA positive or HCV-RNA>ULN);
9. History of immunodeficiency, including testing positive for HIV or suffering from other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
10. Participants who were expected to use systemic strong inhibitors of CYP3A4 within 28 days prior to the start of the study drug and/or during the study period, including, but not limited to, atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, or strong inducers of CYP3A4, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's Wort, or strong inducers or inhibitors of p-gp;
11. Participants with a history of other malignancies. This did not include those who were cured of non-melanoma skin cancer, carcinoma in situ of the cervix, or prostate intraepithelial neoplasm. Participants diagnosed with other malignancies more than 5 years before enrollment could be included only if: (i) there were no active lesions, (ii) the Investigator assessed the risk of recurrence as low, and (iii) the condition would not interfere with the assessment of the efficacy of taletrectinib;
12. Participants who, in the Investigator's judgment, had other serious acute or chronic physical illnesses, mental illnesses, or laboratory abnormalities, as well as diseases or abnormalities that might pose an excessive risk in relation to participation in the study or administration of the study drug;
13. Expected to use any other antitumor drugs within 14 days prior to starting the study drug and/or during the study, including traditional Chinese medicines, Chinese patent drugs, and herbal medicines (including decoctions) with clear antitumor indications in the package inserts;
14. Participants with a known history of neurological or psychiatric disorders, such as epilepsy or dementia, that may affect compliance;
15. Participants with a history of drug or substance abuse;
16. Participants with spinal cord compression due to the tumor (unless the participant's pain is fully controlled and neurological function is stable or restored), cancerous meningitis, or leptomeningeal disease; those assessed by the Investigator to be at risk for brain herniation;
17. Participants with active peptic ulcers, significant vomiting, chronic diarrhea, intestinal obstruction, malabsorption, or other known diseases that could affect drug absorption; those with swallowing difficulties or other severe conditions that significantly affect drug absorption, such as those who have undergone gastric or intestinal resection;
18. Participants with a history or current conditions within 3 months prior to enrollment: heart failure (New York Heart Association functional classification ≥3), myocardial infarction, cerebral infarction, unstable angina, arrhythmias requiring treatment, uncontrollable atrial fibrillation (of any grade), coronary or peripheral artery disease, pulmonary embolism, uncontrollable deep vein thrombosis, or other clinically significant severe thrombosis, or autoimmune diseases requiring treatment; or whose ECG showed a QTc >470 ms (females) or QTc >450 ms (males) before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Approximately 24 months
  Assessed by an Independent Review Committee (IRC) based on the RECIST 1.1 criteria or the RANO criteria.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 24 months
  Assessed by the Investigator based on RECIST 1.1 or RANO criteria.
Duration of response (DOR) | Approximately 24 months
  Assessed separately by the IRC and the Investigator based on RECIST 1.1 or RANO criteria.
Time to Response (TTR) | Approximately 24 months
  Assessed separately by the IRC and the Investigator based on RECIST 1.1 or RANO criteria
Time to Progress (TTP) | Approximately 24 months
  Assessed separately by the IRC and the Investigator based on RECIST 1.1 or RANO criteria.
Disease control rate (DCR) | Approximately 24 months
  Assessed separately by the IRC and the Investigator based on RECIST 1.1 or RANO criteria.
Intracranial objective response rate (IC-ORR) | Approximately 24 months
  Assessed by the IRC based on the RANO-BM criteria for participants with brain metastases at baseline.
Intracranial duration of response (IC-DOR) | Approximately 24 months
  Assessed by the IRC based on the RANO-BM criteria for participants with brain metastases at baseline.
Intracranial disease control rate (IC-DCR) | Approximately 24 months
  Assessed by the IRC based on the RANO-BM criteria for participants with brain metastases at baseline.
Progression free Survival (PFS) | Approximately 30 months
  Progression free Survival (PFS) as assessed separately by the IRC and the Investigator based on RECIST 1.1 or RANO criteria.
Overall survival (OS) | Approximately 36 months
  Assessed by Kaplan-Meier method.
Safety and tolerability of taletrectinib treatment | Approximately 36 months
  Adverse events (AEs)/Serious adverse events (SAEs)/Adverse events of special interests (AESIs); laboratory tests, vital signs, physical examination, ophthalmological examination, 12-lead electrocardiogram (ECG), etc.
Pharmacokinetics (PK) of taletrectinib | Cycle 1 Day 1 to Cycle 2 Day 1
  Plasma concentrations of taletrectinib (in free form)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No